CLINICAL TRIAL: NCT06425848
Title: Hemodynamic Frontiers in Heart Failure Registry
Brief Title: HF2 Registry - Hemodynamic Frontiers in Heart Failure Registry
Acronym: HF2 Registry
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00147383
Record Dates: First submitted 2024-02-29; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure
Keywords: Pulmonary Artery (PA) pressure monitor
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Retrospective arm: Patients who underwent PA pressure implantation from January 1, 2019 will be identified for registry participation. Patients who were implanted before November 8, 2022 will be considered enrolled in the retrospective arm of the registry and may not need to consent if consent waiver is granted by the institutional IRB (Institutional Review Board).
  Interventions: Device: Observational
- Prospective arm: Patients will be identified as eligible for PA pressure sensor implant by a heart failure cardiologist. Patients will consent for device implant and procedure (right heart catheterization) as per standard of care. Patients may also consent to registry participation as per local institutional guidelines and requirements.
  Interventions: Device: Observational

INTERVENTIONS:
Device: Observational — We are collecting information for both retrospective and prospective arm to further understand the utility of PA pressure sensors.

SUMMARY:
The purpose of the HF2 (Hemodynamic Frontiers in Heart Failure) registry is to collect relevant patient-level demographic, clinical, laboratory, and hemodynamic data from patients implanted with pulmonary artery pressure sensor at participating centers to advance scientific knowledge about ambulatory hemodynamics monitoring and HF (Heart Failure) therapies. The data collected will be used for retrospective studies, quality improvement, identifying research cohorts, and member-initiated research.

DETAILED DESCRIPTION:
Longitudinal, multi-center, and non-interventional registry. Patients will be identified as eligible for pulmonary artery pressure sensor implant by a heart failure cardiologist from the heart failure clinic. They will consent for device implant and procedure (right heart catheterization) per standard of care. Patients may also consent to the registry participation, which is optional. They will be informed that the registry intends to gather data and that they may be approached in the future for additional research based on their data and clinical situation. Additionally, patients who underwent pulmonary artery pressure sensor implantation from January 1, 2019, will be identified and consent will be obtained for registry participation, which is optional.

ELIGIBILITY:
Inclusion Criteria:

1. All patients would have been or will be implanted per indications from FDA approval/CHAMPION trial. These would be patients with NYHA (New York Heart Association) Class III heart failure who had a prior hospitalization.
2. Patients who meet the expanded FDA indication (BNP elevation without hospitalization or NYHA class II).

Exclusion Criteria:

1. Patients less than 18 years of age.
2. Pregnant women at the scheduled time of PA pressure sensor implant.
3. Patients unable or unwilling to have continuity of care in the heart failure clinic.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been or will be implanted with PA pressure sensor.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in hemodynamics | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant.
  Hemodynamic data such as mean PA pressure in mmHg, PA systolic pressure in mmHg, PA diastolic pressures in mmHg, will be collected at the time of implant of PA pressure sensor and at 3 months, 6 months, 12 months, 24 months and 36 months post implant.
Changes in Echocardiogram (ECHO) | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  Echo data such as Left Ventricular Ejection Fraction (LVEF) percentage will be collected at implant and at 3 months, 6 months, 12 months, 24 months and 36 months if available.
Medication changes | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  Medications changes such as type of diuretics, will be collected after implant and at 3 months, 6 months, 12 month, 24 months and 36 months. We are not collecting any doses or frequencies.
Sodium | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  Sodium levels, reported as millimoles per liter (mmol/L), will be collected at implant and 3 months, 6 months, 12 months, 24 months and 36 months post implant.
Potassium | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  Potassium level, reported as milliequivalents per liter (mEq/L), will be collected at implant and 3 months, 6 months, 12 months, 24 months and 36 months post implant.
Hemoglobin | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  Hemoglobin concentration (Hb) reported as grams of hemoglobin per deciliter of blood (g/dL). Labs will be collected at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
B-type natriuretic peptide (BNP) | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  BNP level, reported as 100 picograms per milliliter (pg/mL), will be collected at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
aminoterminal pro B-type natriuretic peptide (NT-proBNP) | at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant
  NT-proBNP level, reported as 100 picograms per milliliter (pg/mL), will be collected at implant, 3 months, 6 months, 12 months, 24 months and 36 months post implant

CONTACTS AND LOCATIONS:
Overall Officials: Hirak Shah, MD, Principal Investigator — University of Kansas Medical Center
Locations (12):
- United States (12):
  - Scripps Health, La Jolla, California
  - Indiana University, Bloomington, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Fairview Health, Maplewood, Minnesota
  - Minneapolis Heart Institute Foundation/ Allina Health, Minneapolis, Minnesota
  - Saint Luke's Health System, Kansas City, Missouri
  - University of North Carolina/ Rex Hospital, Inc., Raleigh, North Carolina
  - Providence Heart Institute, Portland, Oregon
  - Prisma Health, Columbia, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - Austin Heart, Austin, Texas
  - Houston Methodist DeBakey Heart and Vascular Center, Houston, Texas